CLINICAL TRIAL: NCT05053152
Title: A Phase II Double-Blinded, Placebo-Controlled Trial of PROstate OligoMETastatic RadiotHErapy With or Without ANdrogen Deprivation Therapy in Oligometastatic Prostate Cancer (NRG Promethean)
Brief Title: Testing the Addition of the Drug Relugolix to the Usual Radiation Therapy for Advanced-Stage Prostate Cancer, The NRG Promethean Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NRG-GU011; NCI-2021-09164 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GU011 (Other: NRG Oncology); NRG-GU011 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Oligometastatic Prostate Carcinoma; Prostate Adenocarcinoma; Prostate Ductal Adenocarcinoma; Prostate Intraductal Carcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; fluciclovine F-18; Magnetic Resonance Spectroscopy; Glutamate Carboxypeptidase II; relugolix; Radiosurgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (placebo, SABR) (Placebo Comparator): Patients receive placebo PO QD on days 1-180 and undergo SABR for 1-3 weeks in the absence of disease progression or unacceptable toxicity. Patients may also undergo bone scan, CT, MRI, PSMA PET/CT or PET/MRI, and/or fluciclovine F18 PET/CT or PET/MRI at time of disease progression. Patients may optionally undergo urine and blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Other: Fluciclovine F18; Procedure: Magnetic Resonance Imaging; Drug: Placebo Administration; Procedure: Positron Emission Tomography; Procedure: PSMA PET Scan; Radiation: Stereotactic Body Radiation Therapy
- Arm II (relugolix, SABR) (Experimental): Patients receive relugolix PO QD on days 1-180 and undergo SABR for 1-3 weeks in the absence of disease progression or unacceptable toxicity. Patients may also undergo bone scan, CT, MRI, PSMA PET/CT or PET/MRI, and/or fluciclovine F18 PET/CT or PET/MRI at time of disease progression. Patients may optionally undergo urine and blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Other: Fluciclovine F18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: PSMA PET Scan; Drug: Relugolix; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo urine and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT and/or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Fluciclovine F18 — Given fluciclovine F18
  Other Names: (18F)Fluciclovine; (18F)GE-148; 18F-Fluciclovine; [18F]FACBC; Anti-(18f)FABC; Anti-1-Amino-3-[18F]Fluorocyclobutane-1-Carboxylic Acid; Anti-[18F] FACBC; Axumin; Fluciclovine (18F); FLUCICLOVINE F-18; GE-148 (18F); GE-148 F-18
Procedure: Magnetic Resonance Imaging — Undergo MRI and/or PET/MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Placebo Administration — Given PO
  Arms: Arm I (placebo, SABR)
Procedure: Positron Emission Tomography — Undergo PET/CT and/or PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: PSMA PET Scan — Undergo PSMA PET/CT or PET/MRI
  Other Names: Prostate-specific Membrane Antigen PET; PSMA PET; PSMA-Positron emission tomography
Drug: Relugolix — Given PO
  Other Names: N-(4-(1-((2,6-Difluorophenyl)methyl)-5-((dimethylamino)methyl)-1,2,3,4-tetrahydro-3-(6-methoxy-3-pyridazinyl)-2,4-dioxothieno(2,3-d)pyrimidin-6-yl)phenyl)-N'-methoxyurea; Orgovyx; Relumina; TAK 385; TAK-385; TAK385
  Arms: Arm II (relugolix, SABR)
Radiation: Stereotactic Body Radiation Therapy — Undergo SABR
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase II trial compares the usual treatment of radiation therapy alone to using the study drug, relugolix, plus the usual radiation therapy in patients with castration-sensitive prostate cancer that has spread to limited other parts of the body (oligometastatic). Relugolix is in a class of medications called gonadotropin-releasing hormone (GnRH) receptor antagonists. It works by decreasing the amount of testosterone (a male hormone) produced by the body. It may stop the growth of cancer cells that need testosterone to grow. Radiation therapy uses high-energy x rays or protons to kill tumor cells. The addition of relugolix to the radiation may reduce the chance of oligometastatic prostate cancer spreading further.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare conventional radiological progression-free survival (rPFS) for positron emission tomography (PET)-detected, biochemically recurrent, oligometastatic, castration-sensitive prostate cancer patients treated with stereotactic ablative body radiation therapy (SABR) plus placebo versus (vs.) SABR plus relugolix.

SECONDARY OBJECTIVES:

I. Compare conventional or PET-based radiological progression-free survival (prPFS) between treatment arms.

II. Compare patient-reported sexual and hormonal quality of life as assessed by corresponding Expanded Prostate Cancer Index Composite Short Form (EPIC-26) domains between treatment arms.

III. Compare other measures of quality of life obtained from the European Quality of Life Five Dimension Five Level Scale Questionnaire (EQ5D-5L), European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-30), Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue instruments between the two treatment arms.

IV. Compare time to salvage therapy and time to castration-resistance between treatment arms.

V. Compare local progression (SABR-targeted lesion), biochemical progression, distant metastases, prostate cancer-specific mortality, metastasis-free survival, and overall survival between treatment arms.

VI. Determine adverse events rates and compare rates between the two treatment arms.

EXPLORATORY OBJECTIVE:

I. Evaluate genomic and peripheral tissue and blood markers of treatment response.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive placebo orally (PO) once daily (QD) on days 1-180 and undergo SABR for 1-3 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive relugolix PO QD on days 1-180 and undergo SABR for 1-3 weeks in the absence of disease progression or unacceptable toxicity.

Patients may also undergo bone scan, computed tomography (CT), magnetic resonance imaging (MRI), prostate-specific membrane antigen (PSMA) positron emission tomography (PET)/CT or PET/MRI, and/or fluciclovine F18 PET/CT or PET/MRI at time of disease progression. Patients may optionally undergo urine and blood sample collection throughout the trial.

After completion of study treatment, patients are followed up at 9 and 12 months, subsequently every 6 months to month 60, and then annually thereafter or at the time of progression.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of prostate adenocarcinoma at any anatomical location (for example, prostate, metastatic site), including intraductal or ductal carcinoma, at any time before registration
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 within 180 days prior to registration
* Prior curative-intent treatment to the prostate, by either:

  * External beam and/or brachytherapy to: Prostate alone, prostate and seminal vesicles, prostate and pelvic nodes, or radiation to all three sites
  * Radical prostatectomy alone, radical prostatectomy plus postoperative radiotherapy to the prostate bed, or radical prostatectomy plus postoperative radiotherapy to the pelvic nodes.

    * Note: Patients who have received curative intent with radiation prior to prostatectomy are eligible and should be categorized as RT to Intact Prostate since that was the first curative intent
* Must meet study entry criteria based on the following diagnostic workup within 120 days prior to registration:

  * History and physical examination;
  * Fluciclovine or PSMA PET scan;
  * PET must be combined with either CT or MRI, but a diagnostic CT or MRI reading/interpretation is not required
* 1 - 5 oligometastatic lesions in bone and/or nodal/soft tissue (non-abutting nodes are counted separately) sites on fluciclovine or PSMA PET within 180 days prior to registration and includes at least ONE of the following:

  * Bone - each metastasis is counted (for example, 2 distinct lesions in the right ilium count as 2 oligometastatic lesions)
  * Extrapelvic Nodal/ soft tissue - requires at least one extrapelvic inguinal or a nodal/soft tissue lesion superior to the iliac bifurcation (that is, American Joint Committee on Cancer [AJCC] M1a version 8)
  * Note: Although a patient must have bone and/or extrapelvic disease to be eligible, when counting the number of oligometastatic lesions, each lymph node lesion, whether pelvic or extrapelvic, is counted (for example, 2 distinct lymph nodes in the right external iliac basin count as 2 oligometastatic lesions; one extrapelvic and one pelvic node count as 2 oligometastic lesions, etc)
* Serum total prostate-specific antigen (PSA) =< 10.0 ng/mL that also meets ONE of the following PSA recurrence definitions:

  * If patient has received-radiation therapy to intact prostate, either

    * PSA > post-RT nadir PSA + 2 ng/mL obtained within 180 days prior to registration, or
    * PSA > 0.2 ng/mL with at least two rises from post-treatment nadir with the most recent PSA within 180 days prior to registration
  * If patient has received a radical prostatectomy with or without post-op RT, either

    * Current PSA > 0.2 ng/mL, with a second confirmatory PSA > 0.2 ng/mL, with most recent PSA obtained within 180 days prior to registration, or
    * Two consecutive PSA rises from post-operative nadir, with most recent PSA obtained within 180 days prior to registration
* Must have >= 3 PSA values within the last two years since end of primary treatment or within the last 2 years prior to registration, whichever is less

  * Note: PSA doubling time must be calculated by entering all PSA values since end of primary treatment or within the last 2 years prior to registration (whichever is less) into the PSA Doubling Time Calculator found at MDCalc.com
* Serum total testosterone >= 100 ng/dL within 180 days prior to registration

  * Note: Prior androgen deprivation therapy (other than bilateral orchiectomy) is allowed if discontinued prior to registration and serum total testosterone is >= 100 ng/dL
* Total bilirubin: =< 1.5 x institutional upper limit of normal (ULN) (Note: In subjects with Gilbert's syndrome, if total bilirubin is > 1.5 x ULN, subject is eligible if direct bilirubin is =< 1.5 x ULN) (within 180 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]): =< 2.5 x institutional ULN (within 180 days prior to registration)
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated

  * Note: Known positive test for hepatitis B virus surface antigen (HBV sAg) indicating acute or chronic infection would make the patient ineligible unless the viral load becomes undetectable on suppressive therapy. Patients who are immune to hepatitis B (anti-hepatitis B surface antibody positive) are eligible (e.g. patients immunized against hepatitis B)
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load

  * Note: Known positive test for hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection would make the patient ineligible unless the viral load becomes undetectable on suppressive therapy
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* The patient must agree to use a highly effective contraception (even men with vasectomies) if he is having sex with a woman of childbearing potential or with a woman who is pregnant while on study drug and for 2 weeks following the last dose of study drug
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information

Exclusion Criteria:

* Currently on androgen deprivation or anti-androgen therapy
* Spinal cord compression, or spinal intramedullary, brain, and/or visceral (for example liver, etc.) metastasis

  * Note: Spinal metastases (PET-detected) with epidural extension are eligible if there is > 0.3 cm spatial separation between the gross tumor volume and spinal cord. Lung metastases are eligible
* Biopsy-proven prostatic carcinoma with signet-ring, sarcomatoid, or neuroendocrine features (for example, small cell)
* Prior metastatic or non-metastatic, invasive malignancy (except non metastatic, non-melanomatous skin cancer) unless continuously disease free for >= 3 years
* Prior chemotherapy for prostate cancer or bilateral orchiectomy

  * Note: Prior chemotherapy for a different cancer is allowed if continuously disease-free for >= 3 years
* Prior high dose radiotherapy to a lesion (i.e. oligometastatic recurrence by PET)

  * Note: Lesions included in or near a previously irradiated planning target volume (PTV) are eligible as long as previous delivered dose is estimated to be less than an EQD2 of 50 Gy
* Inability to treat all oligometastatic sites with radiotherapy in the judgement of the investigator
* Intrapelvic lymph nodes as only site of prostate cancer recurrence
* Inability to swallow whole, undivided, unchewed, and uncrushed pills
* Known gastrointestinal disorder affecting oral medication absorption
* Co-morbidity defined as follows:

  * Patients with any comorbidities that would prohibit completion of protocol specified therapy
  * Inflammatory bowel disease in patients in whom abdominopelvic radiotherapy is planned
  * History of congenital long QT syndrome
  * Current severe or unstable angina
  * New York Heart Association functional classification III/IV heart failure (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association functional classification)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Radiological progression-free survival (rPFS) | Time from randomization to the occurrence of radiological progression detected by conventional imaging or death from any cause, assessed up to 5 years
  The rPFS curves will be estimated by the Kaplan-Meier method and compared between the two treatment arms using a one-sided, logrank test stratified by the three randomization factors.

SECONDARY OUTCOMES:
Positron emission tomography (PET)-based radiological progression-free survival | Time from randomization to the occurrence of conventional or PET-based radiological progression or death from any cause, assessed up to 5 years
  Will be estimated by the Kaplan-Meier method and compared between treatments arms by stratified logrank test. Cox regression models will also be fit, adjusted for the stratification factors and other prognostic baseline factors, to estimate hazard ratios, together with 95% confidence intervals.
Metastasis-free survival | From randomization to distant metastases or death from any cause, assessed up to 5 years
  Will be estimated by the Kaplan-Meier method and compared between treatments arms by stratified logrank test. Cox regression models will also be fit, adjusted for the stratification factors and other prognostic baseline factors, to estimate hazard ratios, together with 95% confidence intervals.
Overall survival | From randomization to death from any cause, assessed up to 5 years
  Will be estimated by the Kaplan-Meier method and compared between treatments arms by stratified logrank test. Cox regression models will also be fit, adjusted for the stratification factors and other prognostic baseline factors, to estimate hazard ratios, together with 95% confidence intervals.
Sexual and hormonal quality of life | Up to 5 years from randomization
  Assessed by Expanded Prostate Cancer Index Composite Short Form (EPIC-26).
Quality of life | Up to 5 years from randomization
  Assessed by European Quality of Life Five Dimension Five Level Scale Questionnaire (EQ5D-5L) and European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-30).
Fatigue | Up to 5 years from randomization
  Assessed by Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue short form.
Time from randomization to administration of salvage therapy | Up to 5 years from randomization
  Will be analyzed using competing-risk methods where, in each case, death prior to occurrence of the event in question will be considered a competing risk. (In the case of death from prostate cancer, the competing risk will be non-prostate cancer death.) Cumulative incidence curves will be generated and compared using the Fine-Gray method and sub-distribution hazard ratios (SHRs) will be estimated, along with 95% confidence intervals, to summarize the magnitude of the treatment effect. In addition to Fine-Gray tests, we will estimate cause-specific hazard ratios by treating the competing risk as a censored observation via stratified logrank tests and Cox regression modelling.
Time from randomization to castrate-resistant prostate cancer | Up to 5 years from randomization
  Will be analyzed using competing-risk methods where, in each case, death prior to occurrence of the event in question will be considered a competing risk. (In the case of death from prostate cancer, the competing risk will be non-prostate cancer death.) Cumulative incidence curves will be generated and compared using the Fine-Gray method and SHRs will be estimated, along with 95% confidence intervals, to summarize the magnitude of the treatment effect. In addition to Fine-Gray tests, we will estimate cause-specific hazard ratios by treating the competing risk as a censored observation via stratified logrank tests and Cox regression modelling.
Time from randomization to local progression within a stereotactic ablative body radiation therapy (SABR)-targeted lesion | Up to 5 years from randomization
  Will be analyzed using competing-risk methods where, in each case, death prior to occurrence of the event in question will be considered a competing risk. (In the case of death from prostate cancer, the competing risk will be non-prostate cancer death.) Cumulative incidence curves will be generated and compared using the Fine-Gray method and SHRs will be estimated, along with 95% confidence intervals, to summarize the magnitude of the treatment effect. In addition to Fine-Gray tests, we will estimate cause-specific hazard ratios by treating the competing risk as a censored observation via stratified logrank tests and Cox regression modelling.
Time from randomization to biochemical progression | Up to 5 years from randomization
  Will be analyzed using competing-risk methods where, in each case, death prior to occurrence of the event in question will be considered a competing risk. (In the case of death from prostate cancer, the competing risk will be non-prostate cancer death.) Cumulative incidence curves will be generated and compared using the Fine-Gray method and SHRs will be estimated, along with 95% confidence intervals, to summarize the magnitude of the treatment effect. In addition to Fine-Gray tests, we will estimate cause-specific hazard ratios by treating the competing risk as a censored observation via stratified logrank tests and Cox regression modelling.
Time from randomization to the occurrence of distance metastases | Up to 5 years from randomization
  Will be analyzed using competing-risk methods where, in each case, death prior to occurrence of the event in question will be considered a competing risk. (In the case of death from prostate cancer, the competing risk will be non-prostate cancer death.) Cumulative incidence curves will be generated and compared using the Fine-Gray method and SHRs will be estimated, along with 95% confidence intervals, to summarize the magnitude of the treatment effect. In addition to Fine-Gray tests, we will estimate cause-specific hazard ratios by treating the competing risk as a censored observation via stratified logrank tests and Cox regression modelling.
Time from randomization to death from prostate cancer | Up to 5 years from randomization
  Will be analyzed using competing-risk methods where, in each case, death prior to occurrence of the event in question will be considered a competing risk. (In the case of death from prostate cancer, the competing risk will be non-prostate cancer death.) Cumulative incidence curves will be generated and compared using the Fine-Gray method and SHRs will be estimated, along with 95% confidence intervals, to summarize the magnitude of the treatment effect. In addition to Fine-Gray tests, we will estimate cause-specific hazard ratios by treating the competing risk as a censored observation via stratified logrank tests and Cox regression modelling.

OTHER OUTCOMES:
Genomic, peripheral tissue, and blood biomarkers | Up to 5 years from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Bridget F Koontz, Principal Investigator — NRG Oncology
Locations (239):
- United States (236):
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Marin General Hospital, Greenbrae, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - AdventHealth Celebration, Celebration, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - GenesisCare USA - Lakewood Ranch, Lakewood Rch, Florida
  - AdventHealth Orlando, Orlando, Florida
  - GenesisCare USA - Plantation, Plantation, Florida
  - Moffitt Cancer Center at SouthShore, Ruskin, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Moffitt Cancer Center at Wesley Chapel, Wesley Chapel, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Alton Memorial Hospital, Alton, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Gonzales, Gonzales, Louisiana
  - Mary Bird Perkins Cancer Center - Metairie, Metairie, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Michigan Healthcare Professionals Macomb, Macomb, Michigan
  - Michigan Healthcare Professionals Madison Heights, Madison Heights, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Michigan Healthcare Professionals Troy, Troy, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - East Carolina University, Greenville, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Fox Chase Cancer Center - East Norriton Hospital Outpatient Center, East Norriton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Carolina Regional Cancer Center, Myrtle Beach, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - FHCC at EvergreenHealth, Kirkland, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - FHCC at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (3):
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec